CLINICAL TRIAL: NCT03782116
Title: Randomized Controlled Study of Efficacy of Elitone Device For the Treatment of Mild-Moderate Stress Urinary Incontinence
Brief Title: Stress Incontinence Trial With Elitone Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elidah, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0718
Record Dates: First submitted 2018-08-16; First posted 2018-12-20 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The device looks identical, but the waveform is different. Randomization, programming and recording of which waveform is done by a third party separate from those listed above.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): Elitone Surface electrical stimulation with a treatment waveform (medium frequency modulated at 50Hz)
  Interventions: Device: Transcutaneous electrical stimulation (Elitone)
- Control (Sham Comparator): Elitone Sham surface electrical stimulation at a very low frequency not known to contract muscles.
  Interventions: Device: Transcutaneous electrical stimulation (Elitone)

INTERVENTIONS:
Device: Transcutaneous electrical stimulation (Elitone) — Transcutaneous perineal area electrical stimulation
  Other Names: Elitone

SUMMARY:
This is a randomized controlled study in which subjects are assigned to either a treatment group or a control (sham) group. Pre- and post-study outcome measures evaluate the change in incontinence episodes on women with mild-moderate stress urinary incontinence.

DETAILED DESCRIPTION:
The Elitone device delivers electrical muscle stimulation to pelvic floor muscles through a disposable surface electrode shaped to fit the perineal region. In typical use women self-administer treatment 20 minutes per day, 5x per week, for 6-12 weeks. Elidah is initiating a prospective, randomized clinical study to demonstrate device efficacy. The study expands a similar pilot to 60 subjects, adds a control arm (sham device) and includes additional outcome measures. Like the earlier study, subjects will self-administer treatment over multiple weeks while maintaining daily logs of their treatment and incontinence symptoms. This is a home-use study, which does not require clinic visits. Accordingly, this allows subject recruitment from across US.

ELIGIBILITY:
Inclusion Criteria:

Predominant Mild-moderate stress incontinence symptoms as determined by self-reported typical number of accidents of 1 per 24 hours or more.

Exclusion Criteria:

* Severe incontinence as determined by self-reported >5 accidents in 24-hr period
* Currently pregnant, may be pregnant, attempting to become pregnant, or delivery within previous 6 weeks
* Implanted cardiac device, untreated cardiac arrhythmia or suffer from other heart problems.
* Cancer, epilepsy or cognitive dysfunction
* Vaginal or pelvic surgery within previous 6 months
* Complete denervation of the pelvic floor
* History or symptoms of urinary retention, extra-urethral incontinence, overflow incontinence
* Active urinary tract infection (UTI) or history of recurrent UTIs (more than three in a year)
* Recurrent vaginitis (bacterial/fungal)
* Pelvic pain/painful bladder syndrome
* Underlying neurologic/neuromuscular disorder
* Severe Obesity as defined by BMI >= 35
* Chronic coughing
* Impaired decision making, drug or alcohol dependence, or suicidal thoughts.
* Anyone who lacks the capacity to consent for themselves or who requires a legal representative to give informed consent.

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Yes must identify as female
Enrollment: 87 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide At-Home study, Monroe, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Completed Intervetion
Arm/Group | Treatment | Control
Started | 57 | 30
Completed | 40 | 18
Not Completed | 17 | 12
Not completed — Lost to Follow-up | 11 | 7
Not completed — Withdrawal by Subject | 6 | 5
Period: Included in Analysis
Arm/Group | Treatment | Control
Started | 40 | 18
Completed | 35 | 13
Not Completed | 5 | 5
Not completed — Protocol Violation | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 35 | 13 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (13.3) | 44.7 (7.0) | 47.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 13 | 48
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 35 | 13 | 48
Stress incontinence leaks/day [Mean (Standard Deviation); unit: leaks/day] | 2.81 (1.01) | 2.65 (1.17) | 2.76 (1.05)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Assessed by Percent Reduction in Urinary Incontinence Episodes
Description: The percent reduction in average number of urinary incontinence episodes over 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percent reduction in leaks/day
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 13
percent reduction in leaks/day | 52.8 (36.3) | 7.9 (55.9)

2. Secondary Outcome: Efficacy Assessed by Percent Reduction in Average Pad Weight
Description: The percent reduction of pad weight in a day over the 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage reduction in pad weight
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 13
percentage reduction in pad weight | 38.3 (62.4) | 25.3 (48.8)

3. Secondary Outcome: Efficacy Assessed by Change in Incontinence Quality of Life Questionnaire (I-QOL)
Description: The efficacy assessed by change in Incontinence quality of life questionnaire (I-QOL). It comprises 22 questions, to which the subject provides a numeric response on a 1-5 scale. 1 = not at all , 2 = a little, 3 = moderately, 4 = quite a bit and 5 = extremely. The score is the sum of the numeric responses, which can range from 22 to 110. The lower the value the less times it happens and the better outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Change of score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 13
Change of score on a scale | 20.8 (20.8) | 10.3 (21.8)

4. Secondary Outcome: Pads Per Day
Description: Reduction of number of pads used per day
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage reduction
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 13
percentage reduction | 35.0 (34.1) | 8.2 (59.9)

ADVERSE EVENTS:
Time Frame: Duration of the 12-week study
Description: External elextrical muscle stimulation is a non-significant risk treatment. Accordingly, serious adverse events are not anticipated for a study of this size.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/13
Other Adverse Events (participants affected / at risk) | 1/35 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=35) | Control (N=13)
Transient muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT03782116/Prot_SAP_001.pdf